CLINICAL TRIAL: NCT02256657
Title: Acute Coronary Syndrome Quality Improvement in Kerala (ACS QUIK) Cluster Randomized, Stepped Wedge Multi-center Implementation of a Locally-Developed Quality Improvement Toolkit
Brief Title: Study of a Quality Improvement Toolkit in Kerala, India, Among Hospitals Treating Acute Coronary Syndrome Patients
Acronym: ACS QUIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mark Huffman, Assistant Professor in Preventive Medicine and Medicine-Cardiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ACS QUIK; 1K99HL107749-01A1 (NIH); R00HL107749-03 (NIH)
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Step 1: Toolkit Implemented in Month 4 (Experimental): Quality Improvement Toolkit
  Interventions: Behavioral: Quality Improvement Toolkit
- Step 2: Toolkit Implemented in Month 8 (Experimental): Quality Improvement Toolkit
  Interventions: Behavioral: Quality Improvement Toolkit
- Step 3: Toolkit Implemented in Month 12 (Experimental): Quality Improvement Toolkit
  Interventions: Behavioral: Quality Improvement Toolkit
- Step 4: Toolkit Implemented in Month 16 (Experimental): Quality Improvement Toolkit
  Interventions: Behavioral: Quality Improvement Toolkit
- Step 5: Toolkit Implemented in Month 20 (Experimental): Quality Improvement Toolkit
  Interventions: Behavioral: Quality Improvement Toolkit

INTERVENTIONS:
Behavioral: Quality Improvement Toolkit — The quality improvement toolkit is comprised of standardized admission and discharge checklists, clinical pathways, an audit and feedback mechanism through electronic data capture, and a monthly report used in conjunction with root cause analysis meetings. Quality improvement toolkits are implemented by individual hospitals.

SUMMARY:
The trial assesses the effect on 30-day major adverse cardiovascular event (MACE) rate of using a quality improvement toolkit among hospitals in Kerala, India. The quality improvement toolkit includes standardized admission and discharge sets, clinical pathways and an audit and feedback program.

DETAILED DESCRIPTION:
This study is a cluster randomized, stepped wedge clinical trial assessing implementation and effect of a locally-developed quality improvement toolkit for patients with acute coronary syndrome (ACS) in Kerala, India. Hospitals will be randomized after stratification for size to one of five cohorts. After a four-month baseline period, the quality improvement toolkit will be implemented in all hospitals in cohort 1. Through a one-way crossover design, these hospitals will continue to use the quality improvement toolkit through the end of the trial for all acute coronary syndrome (ACS) patients. Cohorts 2 through 5 will implement the quality improvement toolkit at time points 8, 12, 16, and 20 months respectively, continuing the use of the toolkits from that time forward to the end of the study. The primary outcome is 30-day MACE rates, including death, reinfarction stroke, or major bleeding. Rates will be continuously collected and compared at one interim time point for safety and efficacy. Final analysis compares MACE rates before and after implementation of the quality improvement toolkits, accounting for cluster effects of hospital, cohort and time.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with Acute Coronary Syndrome

Exclusion Criteria:

* Below the Age of 18
* Patient without Acute Coronary Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21374 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
30-Day Major Adverse Cardiovascular Events | 30 Days from Hospital Discharge
  Compared with usual care, to evaluate the effect of a locally-developed, evidence-based health care quality improvement toolkit on 30-day major adverse cardiovascular events (MACE [death, reinfarction stroke, or major bleeding]) in patients admitted with acute coronary syndrome, adjusted for hospital, time, and step.

SECONDARY OUTCOMES:
In-Hospital Medication Rates | 30 Days
  Compared with usual care, to evaluate the effect of a locally-developed, evidence-based health care quality improvement toolkit on in-hospital medication prescription rates.
Discharge Medication Rates | 30 Days
  Compared with usual care, to evaluate the effect of a locally-developed, evidence-based health care quality improvement toolkit on discharge medication prescription rates.
Discharge Advice Relative to Healthy Lifestyles | 30 Days
  Compared with usual care, to evaluate the effect of a locally-developed, evidence-based health care quality improvement toolkit on discharge advice relative to healthy lifestyles.
In-Hospital and 30-Day Expanded MACE | 30 Days
  Compared with usual care, to evaluate the effect of a locally-developed, evidence-based health care quality improvement toolkit on in-hospital and 30-day expanded MACE.
Concordance with locally-defined performance measures and in-hospital and 30-day MACE | 30 Days
  To evaluate the association between concordance with locally-defined performance measures for ACS care and in-hospital and 30-day MACE.
Health Related Quality of Life | 30 Days
  To evaluate health related quality of life in post-ACS patients (30-days) using a translated and validated version of the Seattle Angina Questionnaire (SAQ).
Impoverishing Effects of an ACS Event | 30 Days
  To evaluate individual- and household-level impoverishing effects of an ACS event in the context of the recent implementation of a national government insurance program for families below the poverty line.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Huffman, MD, MPH, Principal Investigator — Northwestern University; PP Mohanan, MD, DM, Study Director — WestFort Hi-Tech Hospital; Doirairaj Prabhakaran, MD, DM, Study Chair — Centre for Chronic Disease Control; Donald Lloyd-Jones, MD, ScM, Study Chair — Northwestern University
Locations (63):
- India (63):
  - Government Medical College Alappuzha, Alappuzha, Kerala
  - Samaritan Hospital, Aluva, Kerala
  - Little Flower Hospital & Research Center, Angamaly, Kerala
  - Baby Memorial Hospital, Calicut, Kerala
  - Government Medical College Kozhikode, Calicut, Kerala
  - Metro International Cardiac Centre, Calicut, Kerala
  - Sree Narayana Institute of Medical Sciences, Chalakka, Kerala
  - Rajah Charitable Medical Trust, Chāvakkād, Kerala
  - KVM Hospital, Cherthala, Kerala
  - Sukapuram Hospital, Edappāl, Kerala
  - Irinjalakuda Co-operative Hospital Limited, Irinjālakuda, Kerala
  - Lal Memorial Hospital, Irinjālakuda, Kerala
  - Koyili Hospital, Kannur, Kerala
  - St. Martin De Porres Hospital, Kannur, Kerala
  - Pariyaram Medical College Hospital, Kannur, Kerala
  - Kannur Medical College Super Specialty Hospital, Kannur, Kerala
  - Lourdes Hospital, Kochi, Kerala
  - Lakshmi Hospital, Kochi, Kerala
  - PVS Memorial Hospital, Kochi, Kerala
  - Lisie Hospital, Kochi, Kerala
  - Indira Ghandi Co-operative Hospital, Kochi, Kerala
  - Amrita Institute of Medical Sciences & Research Center, Kochi, Kerala
  - Malankara Orthodox Syrian Church Medical College Hospital, Kolenchery, Kerala
  - AA Rahim Memorial District Hospital, Kollam, Kerala
  - Bishop Benziger Hospital, Kollam, Kerala
  - Dr. K. Damodaran Memoral Hospital, Kollam, Kerala
  - Holy Cross Hospital, Kollam, Kerala
  - Travancore Medical College, Kollam, Kerala
  - Bharath Cardiovascular Institute, Kottayam, Kerala
  - S.H. Medical Centre Hospital, Kottayam, Kerala
  - Government Medical College Kottayam, Kottayam, Kerala
  - Caritas Hospital, Kottayam, Kerala
  - KMCT Medical College, Kozhikode, Kerala
  - St. Joseph's Hospital, Kōthamangalam, Kerala
  - Malabar Institute of Medical Sciences, Kōttakkal, Kerala
  - C.H. Memorial Hospital, Malappuram, Kerala
  - Palakkad Government District Hospital, Palakkad, Kerala
  - Thangam Hospital, Palakkad, Kerala
  - Lakshmi Hospital, Palakkad, Kerala
  - EMS Memorial Hospital, Perintalmanna, Kerala
  - Ramdas Clinic & Nursing Home, Perintalmanna, Kerala
  - Tellicherry Cooperative Hospital, Thalassery, Kerala
  - SK Hospital, Thiruvananthapuram, Kerala
  - Medical College Thiruvananthapuram, Thiruvananthapuram, Kerala
  - Sree Chitra Institute for Medical Sciences and Technology, Thiruvananthapuram, Kerala
  - Ananthapuri Hospital and Research Institute, Thiruvananthapuram, Kerala
  - Noorul Islam Institute of Medical Science & Research Foundation, Thiruvananthapuram, Kerala
  - Sree Gokulam Medical College & Research Foundation, Thiruvananthapuram, Kerala
  - St. Mary's Hospital, Thodupuzha, Kerala
  - Santhi Nursing Home, Thrissur, Kerala
  - WestFort Hi-Tech Hospital Limited, Thrissur, Kerala
  - Jubilee Mission Medical College & Research Institute, Thrissur, Kerala
  - Elite Mission Hospital, Thrissur, Kerala
  - Mother Hospital Limited, Thrissur, Kerala
  - Aswini Hospital, Thrissur, Kerala
  - Daya General Hospital & Specialty Surgery Centre, Thrissur, Kerala
  - St. James Hospital, Thrissur, Kerala
  - Amala Institute of Medical Sciences, Thrissur, Kerala
  - Government Medical College Thrissur, Thrissur, Kerala
  - Modern Hospital, Thrissur, Kerala
  - Pushpagiri Institute of Medical Sciences and Research Centre, Tiruvalla, Kerala
  - PRS Hospital, Trivandrum, Kerala
  - Kerala Institute of Medical Sciences, Trivandrum, Kerala

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for ACS QUIK will be shared through NHBLI BIOLINCC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data have been distributed to NHLBI BIOLINCC.
Access Criteria: Access to data will be managed through NLHBI BIOLINCC request process.

REFERENCES:
- [Background] Huffman MD, Mohanan PP, Devarajan R, Baldridge AS, Kondal D, Zhao L, Ali M, Lloyd-Jones DM, Prabhakaran D. Acute coronary syndrome quality improvement in Kerala (ACS QUIK): Rationale and design for a cluster-randomized stepped-wedge trial. Am Heart J. 2017 Mar;185:154-160. doi: 10.1016/j.ahj.2016.10.026. Epub 2016 Dec 21. PMID 28267469
- [Result] Huffman MD, Mohanan PP, Devarajan R, Baldridge AS, Kondal D, Zhao L, Ali M, Krishnan MN, Natesan S, Gopinath R, Viswanathan S, Stigi J, Joseph J, Chozhakkat S, Lloyd-Jones DM, Prabhakaran D; Acute Coronary Syndrome Quality Improvement in Kerala (ACS QUIK) Investigators. Effect of a Quality Improvement Intervention on Clinical Outcomes in Patients in India With Acute Myocardial Infarction: The ACS QUIK Randomized Clinical Trial. JAMA. 2018 Feb 13;319(6):567-578. doi: 10.1001/jama.2017.21906. PMID 29450524
- [Derived] Pei J, Wang X, Xing Z, Chen P, Su W, Deng S, Hu X. Association between admission systolic blood pressure and major adverse cardiovascular events in patients with acute myocardial infarction. PLoS One. 2020 Jun 19;15(6):e0234935. doi: 10.1371/journal.pone.0234935. eCollection 2020. PMID 32559257
- [Derived] Huffman MD, Mohanan PP, Devarajan R, Baldridge AS, Kondal D, Zhao L, Ali M, Spertus JA, Chan PS, Natesan S, Abdullakutty J, Krishnan MN, Tp A, Renga S, Punnoose E, Unni G, Prabhakaran D, Lloyd-Jones DM; ACS QUIK Investigators. Health-Related Quality of Life at 30 Days Among Indian Patients With Acute Myocardial Infarction. Circ Cardiovasc Qual Outcomes. 2019 Feb;12(2):e004980. doi: 10.1161/CIRCOUTCOMES.118.004980. PMID 30755027
- [Derived] Singh K, Devarajan R, Mohanan PP, Baldridge AS, Kondal D, Victorson DE, Karmali KN, Zhao L, Lloyd-Jones DM, Prabhakaran D, Goenka S, Huffman MD; ACS QUIK Investigators. Implementation and acceptability of a heart attack quality improvement intervention in India: a mixed methods analysis of the ACS QUIK trial. Implement Sci. 2019 Feb 6;14(1):12. doi: 10.1186/s13012-019-0857-7. PMID 30728053
- [Derived] Sarma S, Harikrishnan S, Baldridge AS, Devarajan R, Mehta A, Selvaraj S, Ali MK, Mohanan PP, Prabhakaran D, Huffman MD. Availability, Sales, and Affordability of Tobacco Cessation Medicines in Kerala, India. Circ Cardiovasc Qual Outcomes. 2017 Nov;10(11):e004108. doi: 10.1161/CIRCOUTCOMES.117.004108. PMID 29150536